CLINICAL TRIAL: NCT00003232
Title: Randomized Placebo-Controlled Trial of Mitoxantrone/Prednisone and Clodronate Versus Mitoxantrone/Prednisone Alone in Patients With Hormone Refractory Metastatic Prostate Cancer and Pain
Brief Title: Combination Chemotherapy in Treating Pain in Hormone Refractory Metastatic Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR6; CAN-NCIC-PR6 (Other: PDQ); CDR0000066102 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-04-09 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Pain; Prostate Cancer; Quality of Life
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; pain; quality of life
MeSH Terms: conditions — Pain; Prostatic Neoplasms | interventions — Clodronic Acid; Mitoxantrone; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: clodronate disodium
Drug: mitoxantrone hydrochloride
Drug: prednisone
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Some drugs used in chemotherapy can reduce the pain experienced by some people with cancer. Combining more than one drug may be more effective at reducing cancer pain. It is not known whether receiving combination chemotherapy with clodronate is more effective than receiving combination chemotherapy without clodronate for hormone refractory metastatic prostate cancer.

PURPOSE: Randomized double-blinded phase III trial to compare the effectiveness of combination chemotherapy using mitoxantrone plus prednisone with or without clodronate in treating pain in patients with hormone refractory metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effect of mitoxantrone and prednisone with or without clodronate on localized bone pain in patients with hormone refractory metastatic prostate cancer. II. Compare the overall survival and quality of life of these patients after these treatments.

OUTLINE: This is a randomized, double blinded, placebo controlled, multicenter study. Patients are stratified according to quality of pain (mild vs moderate) and previous corticosteroids or one regimen of non-anthracycline-containing cytotoxic chemotherapy (e.g., estramustine) vs none. Patients are assigned to 1 of 2 treatment arms. Arm I consists of oral prednisone twice a day and intravenous mitoxantrone followed by intravenous clodronate administered over 3 hours every 3 weeks. Arm II consists of oral prednisone twice a day and intravenous mitoxantrone followed by intravenous placebo administered over 3 hours every 3 weeks. Doses are adjusted for myelosuppression. Treatment continues until disease progression (although patients initially on placebo can continue on open-label clodronate) or until the maximum cumulative dose of mitoxantrone is reached. Patients with a palliative response may continue on prednisone and the study drug (clodronate or placebo) until disease progression. Quality of life is assessed before and every 3 weeks during study treatment. A daily pain diary is also maintained. All patients are followed at 2 weeks and then every 3 months until death.

PROJECTED ACCRUAL: This study will accrue 204 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the prostate or metastatic carcinoma of presumptive prostate origin as manifest by the presence of sclerotic bony metastases and a serum PSA level greater than the upper limit of normal Radiologically proven progressive bone disease (e.g., new bone scan lesions, increased uptake of isotope at previous sites of disease, and/or increasing bone pain) Hormone refractory disease (i.e., disease progression or recurrence despite documented castrate levels of serum testosterone achieved by bilateral orchiectomy or antiandrogen therapy) Bone pain due to metastatic disease Patients must have achieved stable analgesia for at least 7 days No uncontrolled epidural metastases

PATIENT CHARACTERISTICS: Age: Any age Performance status: ECOG 0-3 Life expectancy: At least 3 months Hematopoietic: WBC at least 3,000/mm3 Absolute granulocyte count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 3.15 mg/dL Renal: Creatinine less than 2.26 mg/dL Serum calcium no greater than 3.1 mmol/L Cardiovascular: Patients with history of angina pectoris, previous cardiac infarction, hypertension, or valvular or congenital heart disease must have baseline measurement of LVEF exceeding 50% Other: No other malignancy within 5 years except nonmelanomatous skin cancer No active infection or any other contraindication to chemotherapy with mitoxantrone No spinal cord or nerve root compression No unstabilized impending pathological fractures

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: One previous course of chemotherapy allowed No prior mitoxantrone or other anthracycline Endocrine therapy: See Disease Characteristics At least 4 weeks since prior nonsteroidal antiandrogens Radiotherapy: At least 4 weeks since prior radiotherapy At least 8 weeks since prior strontium-89 or samarium-153 Surgery: Not specified Other: No prior bisphosphonate therapy

Max Age: 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 1997-11-24 (Actual); Primary Completion 2002-05-01 (Actual); Study Completion 2009-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald S. Ernst, MD, FRCPC, Study Chair — Tom Baker Cancer Centre - Calgary
Locations (21):
- Canada (21):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Penticton Regional Hospital, Penticton, British Columbia
  - British Columbia Cancer Agency - Fraser Valley Cancer Centre, Surrey, British Columbia
  - B.C. Cancer Agency, Vancouver, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Ottawa Regional Cancer Center - General Division, Ottawa, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Hotel Dieu Hospital - St. Catharines, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Queen Elizabeth Hospital, PEI, Charlottetown, Prince Edward Island
  - McGill University Department of Oncology, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Taylor SK, Ding K, Ernst SD, et al.: Palliative response measurement in a phase III study of patients with prostate cancer and painful bone metastases: secondary analysis of NCIC-CTG PR6. [Abstract] J Clin Oncol 26 (Suppl 15): A-9636, 2008.
- [Result] Ernst DS, Tannock IF, Winquist EW, Venner PM, Reyno L, Moore MJ, Chi K, Ding K, Elliott C, Parulekar W. Randomized, double-blind, controlled trial of mitoxantrone/prednisone and clodronate versus mitoxantrone/prednisone and placebo in patients with hormone-refractory prostate cancer and pain. J Clin Oncol. 2003 Sep 1;21(17):3335-42. doi: 10.1200/JCO.2003.03.042. PMID 12947070
- [Result] Ernst DS, Tannock IF, Venner PM, et al.: Randomized placebo controlled trial of mitoxantrone/prednisone and clodronate versus mitoxantrone/prednisone alone in patients with hormone refractory prostate cancer (HRPC) and pain: National Cancer Insititute of Canada Clinical Trials Group study. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-705, 2002.
- [Derived] Jakob T, Tesfamariam YM, Macherey S, Kuhr K, Adams A, Monsef I, Heidenreich A, Skoetz N. Bisphosphonates or RANK-ligand-inhibitors for men with prostate cancer and bone metastases: a network meta-analysis. Cochrane Database Syst Rev. 2020 Dec 3;12(12):CD013020. doi: 10.1002/14651858.CD013020.pub2. PMID 33270906